CLINICAL TRIAL: NCT07118215
Title: A Phase 1, 3-part, Open-label Study to Evaluate the Effects of KarXT Administration on the Pharmacokinetics of Midazolam, Fexofenadine, and Digoxin in Healthy Adult Participants
Brief Title: A Study to Evaluate the Effects of KarXT on the Drug Levels of Midazolam, Fexofenadine, and Digoxin
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Karuna Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CN012-0013
Record Dates: First submitted 2025-08-05; First posted 2025-08-12 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteer; Pharmacokinetics; BMS-986510; KarXT; Cobenfy; Midazolam; Fexofenadine; Digoxin; Drug-drug interaction
MeSH Terms: interventions — xanomeline; trospium chloride; Midazolam; fexofenadine; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Part 1 (Experimental)
  Interventions: Drug: KarXT; Drug: Midazolam
- Part 2 (Experimental)
  Interventions: Drug: KarXT; Drug: Fexofenadine
- Part 3 (Experimental)
  Interventions: Drug: KarXT; Drug: Digoxin

INTERVENTIONS:
Drug: KarXT — Specified dose on specified days
  Other Names: BMS-986510; Xanomeline; Trospium Chloride
Drug: Midazolam — Specified dose on specified days
  Arms: Part 1
Drug: Fexofenadine — Specified dose on specified days
  Arms: Part 2
Drug: Digoxin — Specified dose on specified days
  Arms: Part 3

SUMMARY:
The purpose of this study is to evaluate the effects of KarXT administration on the drug levels of midazolam, fexofenadine, and digoxin in healthy adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be healthy male and female (INOCBP) as determined by no clinically significant deviation from normal in medical history, physical examination, 12-lead ECG, VS, and clinical laboratory determinations.
* Participants must have BMI of 18.0 to 32.0 kg/m2.

Exclusion Criteria:

* Participants must not have organ dysfunction or any clinically significant deviation from normal in physical examination, VS, ECG, or clinical laboratory determinations beyond what is consistent with the target population reference ranges.
* Participants must not have cirrhosis, biliary duct abnormalities, hepatobiliary carcinoma, and/or active hepatic viral infections based on the LFT results.
* Participants must not have any other significant acute or chronic medical illness, as assessed by the investigator.
* Participants must not have history or high risk of urinary retention, gastric retention, or narrow-angle glaucoma or known history of prostate hypertrophy or nocturia.
* Participants must not have current or recent (within 3 months of first study intervention administration) GI disease that could possibly affect drug ADME (eg, bariatric procedure).
* Participants must not have any major surgery, including GI surgery (eg, cholecystectomy and any other GI surgery) that could impact upon the absorption of study intervention (uncomplicated appendectomy and hernia repair are acceptable).
* Participants must not have history of active GI obstructive disorder.
* Participants must not have history of bladder stones.
* Participants must not have history of recurrent urinary tract infections.
* Other protocol define inclusion/exclusion criteria apply.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2026-04-05 (Estimated); Study Completion 2026-04-05 (Estimated)

PRIMARY OUTCOMES:
Part 1: Geometric mean ratio (GMR) of Maximum observed plasma concentration (Cmax) of midazolam with and without KarXT | Up to approximately day 24
Part 1: GMR of Area under the plasma concentration-time curve (AUC) of midazolam with and without KarXT | Up to approximately day 24
Part 2: GMR of Cmax of fexofenadine with and without KarXT | Up to approximately day 24
Part 2: GMR of AUC of fexofenadine with and without KarXT | Up to approximately day 24
Part 3: GMR of Cmax of digoxin with and without KarXT | Up to approximately day 24
Part 3: GMR of AUC of digoxin with and without KarXT | Up to approximately day 24

SECONDARY OUTCOMES:
Number of participants wtih adverse events (AEs) | Up to approximately day 47
  Part 1, 2 and 3
Number of participants wtih serious adverse events (SAEs) | Up to approximately day 47
  Part 1, 2 and 3
Number of participants with physical examination abnormalities | Up to approximately day 24
  Part 1, 2 and 3
Number of participants with vital sign abnormalities | Up to approximately day 24
  Part 1, 2 and 3
Number of participants with 12-lead electrocardiogram abnormalities (ECGs) | Up to approximately day 24
  Part 1, 2 and 3
Number of participants with clinical laboratory assessment abnormalities | Up to approximately day 24
  Part 1, 2 and 3
Number of participants with suicidal ideation with the use of the Columbia-Suicide Severity Rating Scale (C-SSRS) | Up to approximately day 24
  Part 1, 2 and 3
Number of participants with adverse event of special interest (AESIs) | Up to approximately day 47

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- ICON - Lenexa, Lenexa, Kansas, United States

IPD SHARING:
Plan to Share IPD: Yes
BMS will provide access to individual anonymized participant data upon request from qualified researchers, and subject to certain criteria.
  Additional information regarding Bristol Myer Squibb's data sharing policy and process can be found at:
  https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosurecommitment.html
Supporting Information: Study Protocol, SAP, CSR
Time Frame: See Plan Description
Access Criteria: See Plan Description
URL: https://www.bms.com/researchers-and-partners/clinical-trials-and-research/disclosure-commitment.html

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsclinicaltrials.com/us/en/clinical-trials/NCT07118215.html